CLINICAL TRIAL: NCT00451074
Title: A Six Month Randomized, Clinical Trial of Gentamicin in Duchenne Muscular Dystrophy Subjects With Stop Codon Mutations
Brief Title: Six Month Study of Gentamicin in Duchenne Muscular Dystrophy With Stop Codons
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jerry R. Mendell, Director, Center for Gene Therapy, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS043186; 7R01NS043186 (NIH)
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Stop codon mutations
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gentamicin infusions twice a week for six months — Gentamicin infusions twice a week

SUMMARY:
The purpose of this study is to determine the safety of giving intravenous (IV) gentamicin to boys with Duchenne muscular dystrophy who have stop codon mutations.

DETAILED DESCRIPTION:
The primary purpose of this second cohort is to see if the IV Medication, gentamicin, is safe to give twice a week for six months to boys with Duchenne muscular dystrophy (DMD). Secondarily, we want to know if gentamicin can help strengthen the muscles of boys with DMD who have a particular type of genetic mutation known as a stop codon. The gentamicin is thought to allow for "read-through" of this type of mutation which would allow for the production of dystrophin, a protein which is lacking in boys with DMD.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-20 years
* Duchenne muscular dystrophy documented by written report of stop codon mutation analysis of the dystrophin gene.
* Subject is capable of cooperating for efficacy and safety testing
* Absent dystrophin on muscle biopsy
* Subjects may be untreated, taking prednisone or comparable corticosteroids
* Subjects taking corticosteroids must be on the same dose for at least 3 months (90 days) prior to the start of the study.

Exclusion Criteria:

* Known allergy to any aminoglycoside or sulfate compounds
* Current use of potential nephrotoxic or ototoxic drug
* Current use of corticosteroids has not been stable for 3 months (90) days
* Known mutation at nucleotide 1555 in 12S rRNA gene of mitochondrial DNA (predisposes to aminoglycoside hearing loss and commercially available via Athena Diagnostics Lab). This DNA testing (Hearing susceptibility test) will be made available through funding from this grant.
* Inability to hear within the range of 0 to 25 dB in any hearing frequency by pure tone audiometry
* Cystatin C equal to or > 1.4mg/L
* Other medical condition that would impede the conduct of study (e.g., congestive heart failure)

Ages: 5 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
In this phase 1 clinical trial, safety will be measured via gentamicin trough levels, audiology, and renal function tests. These lab tests will remain in the normal range while infusing gentamicin twice a week for 6 month. | 6 months

SECONDARY OUTCOMES:
Determine if gentamicin given over six months improves muscle strength. | 6 months
Determine if gentamicin given over six months increases dystrophin binding at the muscle membrane. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R. Mendell, M.D., Principal Investigator — The Research Institute at Nationwide Children's Hospital/ Nationwide Children's Hospital
Locations (3):
- United States (3):
  - Neuromuscular Research Institute - Scottsdale Healthcare Hopsital at Shea, Scottsdale, Arizona
  - University of Kansas, Kansas City, Kansas
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Result] Malik V, Rodino-Klapac LR, Viollet L, Mendell JR. Aminoglycoside-induced mutation suppression (stop codon readthrough) as a therapeutic strategy for Duchenne muscular dystrophy. Ther Adv Neurol Disord. 2010 Nov;3(6):379-89. doi: 10.1177/1756285610388693. PMID 21179598
- [Result] Malik V, Rodino-Klapac LR, Viollet L, Wall C, King W, Al-Dahhak R, Lewis S, Shilling CJ, Kota J, Serrano-Munuera C, Hayes J, Mahan JD, Campbell KJ, Banwell B, Dasouki M, Watts V, Sivakumar K, Bien-Willner R, Flanigan KM, Sahenk Z, Barohn RJ, Walker CM, Mendell JR. Gentamicin-induced readthrough of stop codons in Duchenne muscular dystrophy. Ann Neurol. 2010 Jun;67(6):771-80. doi: 10.1002/ana.22024. PMID 20517938
- See also: Center for Gene Therapy, The Research Institute at Nationwide Children's Hospital — http://www.nationwidechildrens.org/center-for-gene-therapy